CLINICAL TRIAL: NCT04370236
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Trial of INB03 in the Treatment of Participants With Pulmonary Complications From Coronavirus Disease (COVID-19)
Brief Title: INB03 for the Treatment of Pulmonary Complications From COVID-19
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: Inmune Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INB03-COVID-19_01
Record Dates: First submitted 2020-04-29; First posted 2020-04-30 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: TNF; XPro1595; DN-TNF; cytokine storm; Quellor; Anti-TNF; Anti-TNF therapy; TNF inhibitor; INB03
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — XENP 1595

STUDY DESIGN:
Intervention Model Description: Placebo + Standard of Care vs. INB03 + Standard of Care
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo + Standard of Care (Placebo Comparator): Patients will receive placebo + standard medical care
  Interventions: Drug: Placebo
- INB03 + Standard of Care (Experimental): Patients will receive INB03 + standard medical care
  Interventions: Drug: INB03

INTERVENTIONS:
Drug: INB03 — Patients will receive up to two once per week subcutaneous injections of 1mg/kg INB03
  Other Names: DN-TNF, XPro1595, XENP345, Quellor
  Arms: INB03 + Standard of Care
Drug: Placebo — Patients will receive up to two once per week subcutaneous injections of Placebo
  Arms: Placebo + Standard of Care

SUMMARY:
The purpose of this study is to determine whether XPro1595 can prevent the progression of respiratory complications in COVID19 patients.

DETAILED DESCRIPTION:
The trial is a Phase 2, double-blind, randomized, placebo-controlled clinical trial of INB03 in participants with pulmonary complications due to COVID-19 infection.

Patients with COVID-19 infection and low blood oxygen levels with at least one high risk factor (see below) are eligible to participate in a 40-day study to determine whether INB03 can prevent the progression of pulmonary complications.

Eligible participants will be randomized (1:1) to receive either INB03 + standard of care (SOC) or Placebo + SOC. Participants randomized to INB03 + SOC will receive a 1mg/kg injection of INB03 after randomization. Patients that remain in the hospital 7 days after the first dose will receive a second dose. A final safety visit will occur on Day 70.

ELIGIBILITY:
Inclusion Criteria:

1. Have one or more of the following comorbidities:

   1. Age ≥ 65 years;
   2. Obesity (BMI ≥ 30);
   3. Hypertension (on one or more drugs for treatment of hypertension);
   4. Diabetes (on one or more drugs for Type I or Type II diabetes);
   5. Cardiovascular disease (on one or more drugs for treatment of cardiovascular disease, other than aspirin);
   6. History of congestive heart failure (CHF) or myocardial infarction (MI);
   7. Black or African-American race (at least one parent identifies as Black or African-American);
   8. Hispanic or Latino ethnicity.
2. Have a positive COVID-19 test in the last 28 days;
3. Have room air SaO2 < 96%, or SpO2 < 96% on room air at sea level, or PaO2/FiO2 < 300;
4. Have abnormal chest X-ray, MRI or CT scan consistent with pulmonary complications from COVID-19;
5. Provide written informed consent prior to any study related procedures being performed.

Exclusion Criteria:

Participants will be excluded from the study if 1 or more of the following criteria are applicable at Screening:

1. Age < 18 years;
2. Require immediate intubation due to advanced respiratory failure - including continuous positive airway pressure (CPAP) and bi-level positive airway pressure (BIPAP);
3. Require immediate admission to an Intensive Care Unit (ICU) for any reason;
4. On therapy with approved TNF inhibitor (eg: infliximab, etanercept, adalimumab, certolizumab pegol, golimumab, thalidomide, etc) in the last 6 months;
5. Being treated with dexamethasone (IV or PO) at a dose of >15mg per day or solumedrol or equivalent corticosteroid at a dose of >75mg per day;
6. Taking any medication known to be CCR5 receptor antagonist (eg: leronlimab, aplaviroc, vicriviroc or maraviroc) in the last 6 months;
7. Taking any medication known to inhibit the cytokine pathway (eg: anakinra, tocilizumab, siltuximab, etc) in the last 6 months;
8. Known to be pregnant;
9. Has known HIV, HCV or HBV infection;
10. Has known Mycobacterium tuberculosis infection or evidence of infection on chest X-ray;
11. Significant hepatic disease (ALT/AST> 4 times the ULN);
12. On therapy for cancer in the last 6 months;
13. On therapy for organ transplant in the last 6 months or on a waiting list for organ transplant, including patients on renal replacement therapy for any reason;
14. Known hypersensitivity to investigational product or its excipients;
15. Participating in an investigational drug or device trial;
16. Congestive heart failure (CHF) or myocardial infarction (MI) diagnosed in the last 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with disease progression from randomization to 28 days post-randomization | 28 days
  Disease progression is defined by the development of need for mechanical ventilation or death. Mechanical ventilation includes CPAP, BIPAP or mechanical ventilation requiring intubation.

SECONDARY OUTCOMES:
Proportion of participants with all-cause mortality | 28 days
Proportion of participants who transfer to ICU level care by Day 28 (ICU level care is defined as a hospital setting where patient to nurse ratio is < 4); | 28 days
Proportion of participants with a new onset of neurologic disease (requiring medical intervention), including stroke by Day 28; | 28 days
Proportion of participants with evidence of new CHF or new MI requiring medical intervention by Day 28; | 28 days
Proportion of participants with a new onset embolus or thrombus by Day 28; | 28 days
Proportion of participants who develop a need for renal replacement therapy (defined as need for any type of dialysis including intermittent or continuous peritoneal or hemodialysis) by Day 28; | 28 days
Proportion of participants with an increase in the WHO Ordinal Scale of Clinical Improvement score at any time during the study; | 28 days
Length of hospital stay defined as the number of days in hospital from time of randomization to time of discharge or death, whichever occurs first; | 28 days
Change from baseline in inflammation markers over time. | 28 days

OTHER OUTCOMES:
Incidence of adverse events and serious adverse events not due to underlying disease | 28 days
Incidence of abnormal findings in clinical safety laboratory parameters, vital signs, and ECGs. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tesi, MD, Study Chair — Inmune Bio, Inc.
Locations (9):
- United States (9):
  - NEA Baptist, Jonesboro, Arkansas
  - St. Bernard's, Jonesboro, Arkansas
  - Jewish Hospital, Louisville, Kentucky
  - Mississippi Baptist, Kosciusko, Mississippi
  - Baptist Memorial Hospital-DeSoto, Southard, Missouri
  - Richmond University Medical Center, Staten Island, New York
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - Memorial Hermann, Houston, Texas
  - Memorial Hermann Southeast, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company Website — http://www.inmunebio.com